CLINICAL TRIAL: NCT07388849
Title: Can Rest-Activity Rhythm Profiles Predict Major Depressive Disorder? A Longitudinal Follow-up Study
Brief Title: A Longitudinal Follow-Up Study on Predicting Major Depressive Disorder From Rest-Activity Rhythm Profiles
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Associate Professor, Chinese University of Hong Kong
Other Study IDs: PSY039
Record Dates: First submitted 2026-01-16; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder (MDD); Sleep Disorders; Circadian Rhythm
Keywords: Actigraphy; Major Depressive Disorder; Rest-activity Rhythm; Longitudinal Study
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Major Depressive Disorder Group: This group includes participants who meet the DSM-5 diagnostic criteria for current Major Depressive Disorder based the structured clinical interview SCID-5-RV.
  In this study, all participants will be given a structured clinical interview SCID-5-RV, complete the baseline assessment and then proceed to 14 days of monitoring of sleep, mood, and activity levels. Objective sleep measurements will be collected through actigraphy (e.g., ActiGraph accelerometer), while subjective sleep measurements will be collected using a 14-day sleep diary and self-report measures. The participants who are eligible for actigraphy assessment will also be instructed to wear the device on their non-dominant wrist 24 hours a day for 14 consecutive days.
- Control Group: This group includes participants who do not meet the DSM-5 diagnostic criteria for current Major Depressive Disorder based the structured clinical interview SCID-5-RV.
  In this study, all participants will be given a structured clinical interview SCID-5-RV, complete the baseline assessment and then proceed to 14 days of monitoring of sleep, mood, and activity levels. Objective sleep measurements will be collected through actigraphy (e.g., ActiGraph accelerometer), while subjective sleep measurements will be collected using a 14-day sleep diary and self-report measures. The participants who are eligible for actigraphy assessment will also be instructed to wear the device on their non-dominant wrist 24 hours a day for 14 consecutive days.

SUMMARY:
This proposed study will be a longitudinal follow-up study of a case-control study of 160 participants (CREC Ref: 2023.234). This study aims to follow up on the trajectory of depression and rest-activity rhythm (RAR) disruptions, as well as examine their association over time. The investigators aim to identify distinctive RAR profiles of MDD using the data from the original project and hypothesize that two or more groups will be identified based on individual RAR variables using cluster analysis. The investigators hypothesize that significant differences in depressive symptom severity, sleep quality, and other outcome measures collected in this follow-up will be found between the clustered groups. Individuals exhibiting the most disrupted RAR profiles are hypothesized to have the greatest deterioration in depression symptom severity and other outcome measures. The investigators also hypothesize that people persisting with MDD will exhibit greater disruptions in RAR compared to those without MDD at the follow-up. Furthermore, the investigators will examine whether individual RAR parameters are longitudinally associated with changes in depression symptom severity and other outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 to 70 years
* Chinese language fluency
* Accessibility to an Internet-enabled mobile device
* A willingness to provide informed consent and comply with the study protocol

Exclusion Criteria:

* Severe medical or neurocognitive disorders that make participation unsuitable
* History of electroconvulsive therapy (ECT)
* An unstable use of psychotropic drugs (medication use has to remain stable for at least 6 weeks before baseline assessment)
* Current involvement in any psychological treatment program that targets depression and/or sleep problems
* The investigators will not exclude those with current suicidal risks (i.e., non-fleeting intent or plan), which is a common symptom of MDD. However, if serious suicidal risk (i.e., PHQ-9 Item 9 score > 2) is identified, the participant will be referred to the PI (a clinical psychologist) for further assessment and professional mental health services if deemed necessary.

Exclusion criteria for actigraphy assessment:

* Shift work, pregnancy, work, family, or other commitments that interfere with regular sleep-wake patterns
* Presence of other untreated sleep disorders, including narcolepsy, obstructive sleep apnoea (OSA), and restless leg syndrome (RLS)/periodic leg movement disorder (PLMD) based on the cut-off scores of individual sections in SLEEP-50 (narcolepsy ≥ 7; OSA ≥ 15; RLS/PLMD ≥ 7)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be 160 participants (80 participants with Major Depressive Disorder and 80 age- and gender-matched healthy controls) who participated in a case-control study carried out from 2023 Aug to 2025 Feb in Hong Kong. Those participants will be invited to participate in this study via message, phone call, or email.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Research Version of the Structured Clinical Interview for DSM-5 (SCID-5-RV) | Baseline
  A structured clinical interview for making the major DSM-5 diagnoses. This measure will be used to evaluate the presence of major depressive disorder and other psychiatric conditions, including subtypes of depression.

SECONDARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline, Day 7, Day 14
  A 14-item self-report scale used to measure the symptom severity of anxiety (7-item subscale) and depression (7-item subscale). The minimum score is 0 while maximum socre is 42. Higher scores indicate greater distress.
Change in Insomnia Severity Index (ISI) | Baseline, Day 7, Day 14
  A 7-item self-report scale commonly used to assess the perceived severity of insomnia. The minimum score is 0 while maximum socre is 28. Higher scores indicate greater distress.
Change in the Young Mania Rating Scale (YMRS) | Baseline, Day 7, Day 14
  An 11-item scale used to assess subjective manic symptoms. The minimum score is 0 while maximum socre is 60. Higher scores indicate greater distress.
Change in the Morningness-Eveningness Questionnaire (MEQ) | Baseline, Day 7, Day 14
  A 19-item self-report questionnaire used to measure the chronotype of human circadian rhythms. The minimum score is 16 while maximum socre is 86. Lower scores indicate eveningness, while higher scores indicate morningness.
Change in the Positive and Negative Affect Schedule (PANAS) | 14-day daily survey
  A 20-item scale commonly used to measure positive (10-item subscale) and negative affect (10-item subscale). Each item is rated on a 5-point Likert scale ranging from 1 to 5. Total scores on the scale range from 20 to 100, with higher scores on each subscale indicating greater levels of the respective affect. Specifically, a higher score on the positive affect subscale reflects higher levels of positive emotions, while a higher score on the negative affect subscale reflects higher levels of negative emotions.
Change in the Multidimensional Fatigue Inventory (MFI-20) | Baseline, Day 7, Day 14
  A 20-item scale used to assess five dimensions of fatigue, with each subscale score ranging from 4 to 20. The total score ranges from 20 to 100. Higher scores indicate more severe fatigue.
Change in the Short Form (6-Dimension) Health Survey (SF-6D) | Baseline, Day 7, Day 14
  A health survey used for measuring the quality of life on six dimensions. The scale is scored by converting participants' responses across six health dimensions into predefined utility weights and combining them using a standard multi-attribute algorithm to produce a single health-related quality-of-life score ranging from approximately 0.29 (worst) to 1.00 (full health). Higher scores indicate better health.
Change in sleep time | 14-day daily survey
  Recorded daily using the Consensus Sleep Diary.
Change in wake time | 14-day daily survey
  Recorded daily using the Consensus Sleep Diary.
Change in perceived sleeping quality | 14-day daily survey
  Recorded daily using the Consensus Sleep Diary. The minimum score is 1 while the maximum score is 4. Higher scores indicate better perceived sleeping quality.
Change in use of hypnotics | 14-day daily survey
  Recorded daily using the Consensus Sleep Diary.
Change in actigraphy-derived rest-activity pattern | 14-day on a daily basis, 24 hours a day
  24-hour rest-activity pattern will be collected using research-grade wearables (actigraphy), a validated physiological measurement tool that continuously records movement to estimate sleep-wake cycles. Participants will be instructed to wear the actigraphy on their non- dominant wrist, 24 hours a day, for 14 consecutive days, with exceptions during water sports activities.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong, Hong Kong